CLINICAL TRIAL: NCT03005093
Title: Reliability and Validity of the Turkish Feeding/Swallowing Impact Survey
Brief Title: The Turkish Feeding/Swallowing Impact Survey
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, SELEN SEREL ARSLAN, Principal Investigator, Hacettepe University
Other Study IDs: HACETTEPE UNI
Record Dates: First submitted 2016-12-19; First posted 2016-12-29 (Estimated); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Deglutition Disorder; Dysphagia; Outcome Assessment; Quality of Life
MeSH Terms: conditions — Deglutition Disorders | interventions — Caregivers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- CAREGIVERS: Caregivers of pediatric patients with swallowing disorders will be recruited.
  Interventions: Other: CAREGIVERS
- CHILDREN OF CAREGIVERS: Pediatric patients with swallowing disorders will be recruited.
  Interventions: Other: CHILDREN OF CAREGIVERS

INTERVENTIONS:
Other: CAREGIVERS — The Turkish Feeding/Swallowing Impact Survey will be completed by the caregivers
  Groups: CAREGIVERS
Other: CHILDREN OF CAREGIVERS — Chewing performance with Karaduman Chewing Performance Scale, tongue control with Tongue Thrust Rating Scale, dysphagia symptom severity with the Pediatric version of the Eating Assessment Tool will be evaluated. These assessments will be done before and after swallowing rehabilitation program.
  Groups: CHILDREN OF CAREGIVERS

SUMMARY:
The purpose of this study is to test the reliability and validity of the Turkish Feeding/Swallowing Impact Survey among caregivers of pediatric patients with swallowing disorders.

DETAILED DESCRIPTION:
The purpose of this study is to test the reliability and validity of the Turkish Feeding/Swallowing Impact Survey among caregivers of pediatric patients with swallowing disorders.The internal consistency, test-retest reliability, and criterion validity of T-EAT-10 will be investigated. The internal consistency will be assessed using Cronbach's alpha. Intraclass correlation coefficient (ICC) value with 95 % confidence intervals will be calculated for test-retest reliability. The criterion validity of the scale will be determined by assessing the correlation between the Turkish Feeding/Swallowing Impact Survey and Karaduman Chewing Performance Scale, Tongue Thrust Rating Scale, Pediatric version of the Eating Assessment Tool. The validity will also be determined by completion of the Turkish Feeding/Swallowing Impact Survey before and after swallowing rehabilitation of pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Having a child with swallowing disorders aged between 6 months-18 years

Exclusion Criteria:

* Having a child without swallowing disorders
* Having a child with swallowing disorders aged below 6 months

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Caregivers of pediatric patients with swallowing disorders
Sampling Method: Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2017-01-15 (Actual); Primary Completion 2017-05-15 (Actual); Study Completion 2017-05-15 (Actual)

PRIMARY OUTCOMES:
The Turkish Feeding/Swallowing Impact Survey | 6 months
  This scale is used to determine the concerns of caregivers related to their children feeding/swallowing difficulties

SECONDARY OUTCOMES:
The Karaduman Chewing Performance Scale | 6 months
  This scale is used to determine chewing performance level of children
Tongue Thrust Rating Scale | 6 months
  This scale is used to determine tongue thrust severity of children
Pediatric version of the Eating Assessment Tool | 6 months
  This tool is used to determine initial dysphagia symptom severity of children

CONTACTS AND LOCATIONS:
Overall Officials: SELEN SEREL ARSLAN, PhD, Principal Investigator — Hacettepe University
Locations (1):
- Hacetttepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No